CLINICAL TRIAL: NCT01075152
Title: Trial for the Optimal Timing of HIV Therapy After Cryptococcal Meningitis
Brief Title: Cryptococcal Optimal ART Timing Trial
Acronym: COAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Mbarara University of Science and Technology (Other); Makerere University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0810M49622; U01AI089244 (NIH)
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Cryptococcal Meningitis; HIV Infections; AIDS
Keywords: cryptococcal meningitis; cryptococcus; cryptococcosis; HIV; AIDS; strategy
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; Acquired Immunodeficiency Syndrome; Cryptococcosis | interventions — efavirenz; Nucleosides; Zidovudine; Stavudine; Lamivudine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Earlier HIV Therapy (Experimental): HIV therapy initiated at 7-13 days of cryptococcal meningitis diagnosis. HIV therapy consisting of a nucleoside with lamivudine and efavirenz.
  Interventions: Drug: efavirenz; Biological: nucleoside
- Deferred HIV Therapy (Active Comparator): HIV therapy initiated at 5 weeks after cryptococcal meningitis diagnosis (+/- 1 week).
  HIV therapy consisting of a nucleoside with lamivudine and efavirenz.
  Interventions: Drug: efavirenz; Biological: nucleoside

INTERVENTIONS:
Drug: efavirenz — Treatment strategy of when to initiate first line HIV therapy after cryptococcal meningitis diagnosis.
  Other Names: sustiva
Biological: nucleoside — Treatment strategy of when to initiate first line HIV therapy after cryptococcal meningitis diagnosis.
  Other Names: zidovudine or stavudine; lamivudine

SUMMARY:
The Cryptococcal Optimal ART Timing (COAT) trial seeks to determine after cryptococcal meningitis (CM) whether early initiation of antiretroviral therapy (ART) prior to hospital discharge results in superior survival compared to standard initiation of ART started as an outpatient.

DETAILED DESCRIPTION:
After 7-11 days of amphotericin B therapy, subjects will be randomized in a 1:1 allocation to:

* Early initiation of ART (Experimental Group) = ART initiated within 48 hours after study entry, OR
* Standard initiation of ART (Control Group) = ART at >=4 weeks after study entry

HIV therapy will be with efavirenz plus nucleoside backbone per national guidelines for first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection, documented by ELISA
* Antiretroviral medication naïve (excluding mother-to-child transmission therapy)
* Age >14 years
* Cryptococcal meningitis diagnosed by either culture or CSF cryptococcal antigen (CRAG)
* Ability and willingness of the participant or legal guardian/representative to give informed consent.
* Receiving amphotericin-based anti-fungal therapy

Exclusion Criteria:

* Study entry prior to receipt of <7 days or >11 days of amphotericin therapy
* History of prior, known cryptococcal meningitis
* Inability to take enteral medication
* Receiving chemotherapy or other immunosuppressant medications
* Cannot or unlikely to attend regular clinic visits
* Contraindication to immediate or delayed HIV therapy based on serious co-morbidities or co-infections, or laboratory values
* Pregnancy or Breastfeeding
* Female participants of childbearing potential who are participating in sexual activity that could lead to pregnancy must agree to use two reliable methods of contraception

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Boulware, MD, MPH, Principal Investigator — University of Minnesota
Locations (3):
- GF Jooste Hospital, Cape Town, South Africa
- Uganda (2):
  - Infectious Disease Institute, Mulago Hospital, Makerere University, Kampala
  - Mbarara University of Science and Technology, Mbarara

REFERENCES:
- [Background] Rajasingham R, Williams D, Meya DB, Meintjes G, Boulware DR, Scriven J. Nosocomial drug-resistant bacteremia in 2 cohorts with cryptococcal meningitis, Africa. Emerg Infect Dis. 2014 Apr;20(4):722-4. doi: 10.3201/eid2004.131277. No abstract available. PMID 24655747
- [Background] Carlson RD, Rolfes MA, Birkenkamp KE, Nakasujja N, Rajasingham R, Meya DB, Boulware DR. Predictors of neurocognitive outcomes on antiretroviral therapy after cryptococcal meningitis: a prospective cohort study. Metab Brain Dis. 2014 Jun;29(2):269-279. doi: 10.1007/s11011-013-9476-1. Epub 2014 Jan 9. PMID 24399496
- [Background] Boulware DR, Rolfes MA, Rajasingham R, von Hohenberg M, Qin Z, Taseera K, Schutz C, Kwizera R, Butler EK, Meintjes G, Muzoora C, Bischof JC, Meya DB. Multisite validation of cryptococcal antigen lateral flow assay and quantification by laser thermal contrast. Emerg Infect Dis. 2014 Jan;20(1):45-53. doi: 10.3201/eid2001.130906. PMID 24378231
- [Background] Kabanda T, Siedner MJ, Klausner JD, Muzoora C, Boulware DR. Point-of-care diagnosis and prognostication of cryptococcal meningitis with the cryptococcal antigen lateral flow assay on cerebrospinal fluid. Clin Infect Dis. 2014 Jan;58(1):113-6. doi: 10.1093/cid/cit641. Epub 2013 Sep 24. PMID 24065327
- [Background] Robertson EJ, Najjuka G, Rolfes MA, Akampurira A, Jain N, Anantharanjit J, von Hohenberg M, Tassieri M, Carlsson A, Meya DB, Harrison TS, Fries BC, Boulware DR, Bicanic T. Cryptococcus neoformans ex vivo capsule size is associated with intracranial pressure and host immune response in HIV-associated cryptococcal meningitis. J Infect Dis. 2014 Jan 1;209(1):74-82. doi: 10.1093/infdis/jit435. Epub 2013 Aug 14. PMID 23945372
- [Background] Durski KN, Kuntz KM, Yasukawa K, Virnig BA, Meya DB, Boulware DR. Cost-effective diagnostic checklists for meningitis in resource-limited settings. J Acquir Immune Defic Syndr. 2013 Jul 1;63(3):e101-8. doi: 10.1097/QAI.0b013e31828e1e56. PMID 23466647
- [Background] Rajasingham R, Rolfes MA, Birkenkamp KE, Meya DB, Boulware DR. Cryptococcal meningitis treatment strategies in resource-limited settings: a cost-effectiveness analysis. PLoS Med. 2012;9(9):e1001316. doi: 10.1371/journal.pmed.1001316. Epub 2012 Sep 25. PMID 23055838
- [Background] Rolfes MA, Hullsiek KH, Rhein J, Nabeta HW, Taseera K, Schutz C, Musubire A, Rajasingham R, Williams DA, Thienemann F, Muzoora C, Meintjes G, Meya DB, Boulware DR. The effect of therapeutic lumbar punctures on acute mortality from cryptococcal meningitis. Clin Infect Dis. 2014 Dec 1;59(11):1607-14. doi: 10.1093/cid/ciu596. Epub 2014 Jul 23. PMID 25057102
- [Background] Scriven JE, Rhein J, Hullsiek KH, von Hohenberg M, Linder G, Rolfes MA, Williams DA, Taseera K, Meya DB, Meintjes G, Boulware DR; COAT Team. Early ART After Cryptococcal Meningitis Is Associated With Cerebrospinal Fluid Pleocytosis and Macrophage Activation in a Multisite Randomized Trial. J Infect Dis. 2015 Sep 1;212(5):769-78. doi: 10.1093/infdis/jiv067. Epub 2015 Feb 4. PMID 25651842
- [Background] Williams DA, Kiiza T, Kwizera R, Kiggundu R, Velamakanni S, Meya DB, Rhein J, Boulware DR. Evaluation of fingerstick cryptococcal antigen lateral flow assay in HIV-infected persons: a diagnostic accuracy study. Clin Infect Dis. 2015 Aug 1;61(3):464-7. doi: 10.1093/cid/civ263. Epub 2015 Apr 1. PMID 25838287
- [Background] Rajasingham R, Rhein J, Klammer K, Musubire A, Nabeta H, Akampurira A, Mossel EC, Williams DA, Boxrud DJ, Crabtree MB, Miller BR, Rolfes MA, Tengsupakul S, Andama AO, Meya DB, Boulware DR. Epidemiology of meningitis in an HIV-infected Ugandan cohort. Am J Trop Med Hyg. 2015 Feb;92(2):274-9. doi: 10.4269/ajtmh.14-0452. Epub 2014 Nov 10. PMID 25385864
- [Background] Nabeta HW, Bahr NC, Rhein J, Fossland N, Kiragga AN, Meya DB, Dunlop SJ, Boulware DR. Accuracy of noninvasive intraocular pressure or optic nerve sheath diameter measurements for predicting elevated intracranial pressure in cryptococcal meningitis. Open Forum Infect Dis. 2014 Oct 11;1(3):ofu093. doi: 10.1093/ofid/ofu093. eCollection 2014 Dec. PMID 25734161
- [Background] Meya DB, Okurut S, Zziwa G, Rolfes MA, Kelsey M, Cose S, Joloba M, Naluyima P, Palmer BE, Kambugu A, Mayanja-Kizza H, Bohjanen PR, Eller MA, Wahl SM, Boulware DR, Manabe YC, Janoff EN. Cellular immune activation in cerebrospinal fluid from ugandans with cryptococcal meningitis and immune reconstitution inflammatory syndrome. J Infect Dis. 2015 May 15;211(10):1597-606. doi: 10.1093/infdis/jiu664. Epub 2014 Dec 9. PMID 25492918
- [Background] Bahr NC, Rolfes MA, Musubire A, Nabeta H, Williams DA, Rhein J, Kambugu A, Meya DB, Boulware DR. Standardized electrolyte supplementation and fluid management improves survival during amphotericin therapy for cryptococcal meningitis in resource-limited settings. Open Forum Infect Dis. 2014 Aug 25;1(2):ofu070. doi: 10.1093/ofid/ofu070. eCollection 2014 Sep. PMID 25734140
- [Background] Kwizera R, Nguna J, Kiragga A, Nakavuma J, Rajasingham R, Boulware DR, Meya DB. Performance of cryptococcal antigen lateral flow assay using saliva in Ugandans with CD4 <100. PLoS One. 2014 Jul 31;9(7):e103156. doi: 10.1371/journal.pone.0103156. eCollection 2014. PMID 25078453
- [Result] Boulware DR, Meya DB, Muzoora C, Rolfes MA, Huppler Hullsiek K, Musubire A, Taseera K, Nabeta HW, Schutz C, Williams DA, Rajasingham R, Rhein J, Thienemann F, Lo MW, Nielsen K, Bergemann TL, Kambugu A, Manabe YC, Janoff EN, Bohjanen PR, Meintjes G; COAT Trial Team. Timing of antiretroviral therapy after diagnosis of cryptococcal meningitis. N Engl J Med. 2014 Jun 26;370(26):2487-98. doi: 10.1056/NEJMoa1312884. PMID 24963568
- [Derived] Sadiq A, Kwizera R, Kiiza TK, Ayebare P, Ahimbisibwe C, Ndyetukira JF, Boulware DR, Meya DB. Experiences, challenges, gaps, and strategies for counselling persons presenting with advanced HIV-associated meningitis in Uganda. AIDS Res Ther. 2025 Feb 19;22(1):21. doi: 10.1186/s12981-025-00705-z. PMID 39972326
- [Derived] Kwizera R, Sadiq A, Ndyetukira JF, Nalintya E, Williams D, Rhein J, Boulware DR, Meya DB; COAT and ASTRO trial teams. Impact of community engagement and social support on the outcomes of HIV-related meningitis clinical trials in a resource-limited setting. Res Involv Engagem. 2020 Aug 20;6:49. doi: 10.1186/s40900-020-00228-z. eCollection 2020. PMID 32843994
- [Derived] Skipper C, Schleiss MR, Bangdiwala AS, Hernandez-Alvarado N, Taseera K, Nabeta HW, Musubire AK, Lofgren SM, Wiesner DL, Rhein J, Rajasingham R, Schutz C, Meintjes G, Muzoora C, Meya DB, Boulware DR. Cytomegalovirus Viremia Associated With Increased Mortality in Cryptococcal Meningitis in Sub-Saharan Africa. Clin Infect Dis. 2020 Jul 27;71(3):525-531. doi: 10.1093/cid/ciz864. PMID 31504335
- [Derived] Bayiyana A, Okurut S, Nabatanzi R, Zziwa G, Boulware DR, Lutwama F, Meya D. Longitudinal Changes in Cd4+, Cd8+ T Cell Phenotype and Activation Marker Expression Following Antiretroviral Therapy Initiation among Patients with Cryptococcal Meningitis. J Fungi (Basel). 2019 Jul 17;5(3):63. doi: 10.3390/jof5030063. PMID 31319498
- [Derived] Tugume L, Rhein J, Hullsiek KH, Mpoza E, Kiggundu R, Ssebambulidde K, Schutz C, Taseera K, Williams DA, Abassi M, Muzoora C, Musubire AK, Meintjes G, Meya DB, Boulware DR; COAT and ASTRO-CM teams. HIV-Associated Cryptococcal Meningitis Occurring at Relatively Higher CD4 Counts. J Infect Dis. 2019 Feb 23;219(6):877-883. doi: 10.1093/infdis/jiy602. PMID 30325463
- See also: NIH NIAID FAQ on COAT Trial (Preliminary Results) — http://www.niaid.nih.gov/news/QA/Pages/COATqa.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Earlier HIV Therapy: HIV therapy initiated at 7-13 days after cryptococcal diagnosis
- Deferred HIV Therapy: HIV therapy initiated at 5 weeks after cryptococcal meningitis diagnosis (+/1 week)
Period: Overall Study
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Started | 88 (randomized) | 89 (randomized)
Completed | 87 | 89
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: HIV-infected persons not previously receiving HIV therapy with first episode of cryptococcal meningitis diagnosed by CSF culture and/or CSF cryptococcal antigen testing.
Groups:
- Earlier HIV Therapy: HIV therapy initiated at 7-13 days after cryptococcal meningitis diagnosis.
- Deferred HIV Therapy: HIV therapy initiated at 5 weeks after cryptococcal meningitis diagnosis (+/- 1 week)
- Total: Total of all reporting groups
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy | Total
Number analyzed (Participants) | 88 | 89 | 177
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [28 to 40] | 36 [30 to 40] | 35 [29 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 84
  Male | 46 | 47 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 88 | 89 | 177
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 75 | 77 | 152
  South Africa | 13 | 12 | 25
CD4 Count, baseline [Median (Inter-Quartile Range); unit: cells/mcL] | 19 [9 to 69] | 28 [11 to 76] | 23 [10 to 73]
CSF Quantitative Culture, baseline [Median (Inter-Quartile Range); unit: log10 colony forming units/mL of CSF] | 5.3 [4.2 to 5.7] | 4.8 [3.8 to 5.5] | 5.1 [4.0 to 5.6]
CSF Cryptococcal Antigen titer, 1:xxxx [Median (Inter-Quartile Range); unit: titers] — as performed by serial dilutions with lateral flow assay (LFA)
  titers | 8000 [2000 to 16000] | 4000 [1000 to 14400] | 6400 [2000 to 16000]
HIV-1 Viral Load [Median (Inter-Quartile Range); unit: log10 copies/mL] | 5.5 [5.2 to 5.8] | 5.5 [5.3 to 5.8] | 5.5 [5.2 to 5.8]

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Intention to treat analysis of 26 week survival of all subjects enrolled. Reported below are the numbers of participants who died by Week 26.
Time Frame: 26 weeks from study entry
Measure: Number; unit: participants
Groups:
- Deferred HIV Therapy: HIV therapy initiated at 5 weeks after cryptococcal meningitis (+/- 1 week).
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 88 | 89
participants | 40 | 27
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; We compared the randomization arms for the primary endpoint of survival using time-to-event methods of Cox proportional hazards models by the intention-to-treat principle, based on two-sided type-I error with alpha=0.05. The trial was statistically powered to detect a 25% relative survival benefit (15% absolute benefit) with 90% power and overall two-sided alpha=0.05 with an intended sample size of 500 participants. The trial was halted early by the Data and Safety Monitoring Board; Test type: Superiority or Other; p = 0.03, Regression, Cox — A Lan-DeMets spending function analog of the O'Brien-Fleming boundaries was proposed to control the type-I error resulting from multiple interim analyses; Hazard Ratio (HR) = 1.73, 95% CI 2-sided [1.06 to 2.82] — Hazard Ratio describes the risk of earlier HIV therapy in comparison to deferred HIV therapy initiation as the reference group

2. Secondary Outcome: Incidence of Immune Reconstitution Inflammatory Syndrome
Description: Incidence of cryptococcal-related immune reconstitution inflammatory syndrome through 46 weeks after enrollment.
Time Frame: 46 weeks
Population: analysis is of persons who survived to initiate HIV therapy
Measure: Number; unit: participants
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 87 | 69
participants | 17 | 9
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; To account for the competing risk of death, the cumulative incidence function compared the randomized groups for endpoints of IRIS, relapse, and adverse events (Gray's method); Test type: Superiority or Other; p = 0.32, Gray's method of cumulative incidence

3. Secondary Outcome: Incidence of Cryptococcal-relapse
Description: Incidence of culture positive cryptococcal meningitis relapse
Time Frame: 46 weeks
Measure: Number; unit: participants
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 88 | 89
participants | 2 | 8
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.06, Gray's method of cumulative incidence

4. Secondary Outcome: Safety of ART Initiation
Description: Incidence of Adverse Events (Grade 3,4,5) through 46-weeks, as defined by the National Institute of Allergy and Infectious Diseases, Division of AIDS toxicity classification scale, version 2009.
Time Frame: 46 weeks
Measure: Number; unit: participants
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 88 | 89
participants | 73 | 75
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; Categorical secondary endpoints were compared with Fisher's exact tests; Test type: Superiority or Other; p = 0.98, Fisher Exact

5. Secondary Outcome: 46-week Survival
Description: 46-week survival by time-to-event analysis of all subjects enrolled
Time Frame: 46 weeks
Measure: Number; unit: participants
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 88 | 89
participants | 41 | 29
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; We compared the randomization arms for survival using time-to-event methods of Cox proportional hazards models; Test type: Superiority or Other; p = 0.04, Regression, Cox; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [1.03 to 2.68]

6. Secondary Outcome: HIV-1 Viral Suppression
Description: HIV-1 virologic suppression to <400 copies/mL at 26-weeks after enrollment
Time Frame: 26 weeks
Population: Among persons alive at 26 weeks. 1 participant in the early ART arm had consent withdrawn by their family on day 2 after study entry. 3 participants in the deferred ART arm missing their 26 week viral load sampling.
Measure: Number; unit: participants
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 47 | 59
participants | 43 | 49
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; Categorical secondary endpoints were compared with Fisher's exact tests; Test type: Superiority or Other; p = 0.26, Fisher Exact

7. Secondary Outcome: Antiretroviral Therapy Tolerability
Description: Incidence of antiretroviral therapy interruption by >=3 consecutive days
Time Frame: 26 weeks
Population: Analysis is of persons who survived to initiate HIV therapy.
Measure: Number; unit: participants
Groups:
- Earlier HIV Therapy: HIV therapy initiated at 7-13 days after cryptococcal meningitis diagnosis]
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 87 | 69
participants | 5 | 1
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; Categorical secondary endpoints were compared with Fisher's exact tests; Test type: Superiority or Other; p = 0.23, Fisher Exact

8. Secondary Outcome: Karnofsky Functional Status
Description: Functional status via Karnofsky performance status score at 4, 26, 46 weeks.
  Karnofsky Scale:
  100 - Normal; no complaints; no evidence of disease. 90 - Able to carry on normal activity; minor signs or symptoms of disease. 80 - Normal activity with effort; some signs or symptoms of disease. 70 - Cares for self; unable to carry on normal activity or to do active work. 60 - Requires occasional assistance, but is able to care for most of his personal needs.
  50 - Requires considerable assistance and frequent medical care. 40 - Disabled; requires special care and assistance. 30 - Severely disabled; hospital admission is indicated although death not imminent.
  20 - Very sick; hospital admission necessary; active supportive treatment necessary.
  10 - Moribund; fatal processes progressing rapidly. 0 - Dead
Time Frame: 46 weeks
Population: Analysis is of persons alive at the time point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 88 | 89
Scores on a scale
  4 weeks | 70 (19) | 70 (19)
  26 weeks | 93 (7) | 93 (10)
  46 weeks | 92 (10) | 95 (8)
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; The overall change from baseline in Karnofsky performance status scores was compared between groups via a repeated measure analysis, unstructured covariance matrix, adjusted for baseline value; Test type: Superiority or Other; p = 0.34, repeated measure analysis

9. Secondary Outcome: Microbiologic Clearance
Description: Microbiologic clearance of cryptococcus as measured by serial quantitative cryptococcal cultures collected at diagnosis through 14 days of amphotericin therapy. The early fungicidal activity (EFA) of the rate of clearance is expressed as log10 colony forming units (CFU) of Cryptococcus neoformans per mL of CSF per day.
Time Frame: 4 weeks
Population: All participants with >2 quantitative CSF cultures obtained
Measure: Mean (95% Confidence Interval); unit: log10 CFU/mL/day
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 83 | 83
log10 CFU/mL/day
  EFA by mixed effects model | -0.31 [-0.34 to -0.28] | -0.31 [-0.34 to -0.28]
  EFA by linear regression | -0.39 [-0.45 to -0.32] | -0.35 [-0.39 to -0.31]
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; To describe early fungicidal activity, a linear mixed effects regression model fit with a random intercept and slope estimated the rate of clearance of log10 colony forming units (CFU) of Cryptococcus, per mL of CSF per day, for all participants with >2 cultures obtained; Test type: Superiority or Other; p = 0.44, Regression, Linear; a linear mixed effects regression model fit with a random intercept and slope estimated the rate of clearance

10. Other Pre Specified Outcome: Percentage of Participants, Per CSF WBC Subgroup, Who Died by Week 26
Description: Percentage of Participants who died by week 26 based on CSF white blood cell (WBC) count at study entry (time of randomization at a median of 8 days of anti-fungal therapy).
Time Frame: 26 weeks
Population: among persons with a measured CSF white cell count at randomization (Day 7-11 of amphotericin treatment)
Measure: Number; unit: percentage of participants
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Number analyzed (Participants) | 75 | 71
percentage of participants
  CSF WBC <5 /mcl (n=33, 31) | 48.5 | 16.1
  CSF WBC >5/mcL (n=42, 40) | 40.5 | 45
Statistical Analysis 1: Comparison: Earlier HIV Therapy vs Deferred HIV Therapy; Pre-specified subgroups formed by baseline characteristics were compared for 26 week survival with models including an interaction term between treatment arm and subgroup; Test type: Superiority or Other; p = 0.02, Regression, Cox — This is the interaction p-value for CSF white cell count at randomization (implying there is a statistical difference in the outcome by arm based on this parameter)

ADVERSE EVENTS:
Time Frame: 46 weeks
Description: Grade 3,4,5 adverse events were protocol specified secondary endpoint and were collected.
Arm/Group | Earlier HIV Therapy | Deferred HIV Therapy
Serious Adverse Events (participants affected / at risk) | 49/88 | 53/89
Other Adverse Events (participants affected / at risk) | 73/88 | 75/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Earlier HIV Therapy (N=88) | Deferred HIV Therapy (N=89)
Grade 5 AEs (Nervous system disorders) | 11 (14) | 5 (10) — Death (The number of AEs is greater than the number of persons as multiple AEs could occur simultaneously in the same participant).
Grade 4 Serious AEs (Nervous system disorders) | 38 (59) | 42 (57) — Initial Grade 4 serious AEs
Grade 3 Serious AEs (Nervous system disorders) | 40 (48) | 38 (47) — Grade 3-5 serious AEs
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Earlier HIV Therapy (N=88) | Deferred HIV Therapy (N=89)
Hematology (Blood and lymphatic system disorders) | 41 (99) | 47 (128)
Chemistries (Metabolism and nutrition disorders) | 32 (65) | 25 (53)
Infection (Infections and infestations) | 10 (13) | 18 (26)

LIMITATIONS AND CAVEATS:
The differences in mortality in the two arms were of sufficient magnitude that trial enrollment was stopped early by the Data and Safety Monitoring Board. Historically, trials stopped early routinely over-estimate the magnitude of benefit or harm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No